CLINICAL TRIAL: NCT02475408
Title: Effect of Permanent Internal Mammary Artery Occlusion on Extracardiac Coronary Collateral Supply
Acronym: IMAO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SNCTP000000901
Record Dates: First submitted 2015-01-05; First posted 2015-06-18 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2015-06

CONDITIONS: Circulation, Collateral; Coronary Artery Disease; Internal Mammary-Coronary Artery Anastomosis; Ischemia
Keywords: Circulation, Collateral; Coronary Artery Disease; Internal Mammary-Coronary Artery Anastomosis; Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interventional Study Arm (Experimental): In the presence of a significant right coronary artery stenosis, catheter-based occlusion of the right IMA distal to the take-off of the pericardio-phrenic branch is performed at baseline using a dedicated occlusion device (Amplatzer vascular plug).
  Interventions: Device: Amplatzer vascular plug

INTERVENTIONS:
Device: Amplatzer vascular plug

SUMMARY:
Coronary artery disease and the benefit of bypasses:

Despite considerable advances in medicine, cardiovascular diseases remain the number one cause of death globally, primarily consequence of myocardial infarction (MI). Coronary collaterals exert a protective effect by providing an alternative source of blood flow to a myocardial territory potentially affected by an acute coronary occlusion. Coronary collaterals represent pre-existing inter-arterial anastomoses and as such are the natural counter-part of surgically created bypasses. Sufficient coronary collaterals have been shown to confer a significant benefit in terms of overall mortality and cardiovascular events. In this regard, the concept of augmenting coronary collateral function as an alternative treatment strategy to alter the course of CAD, as well as to control symptoms, is attractive.

Durable promotion of coronary collateral circulation:

Before the advent of coronary artery bypass grafting, permanent augmentation of coronary collateral supply by a single structural modification has already been attempted. Bilateral ligation of the internal mammary arteries (IMA) was performed in CAD patients to alleviate angina pectoris and electrocardiographic (ECG) signs of ischemia. The prevalent in vivo function of natural IMA-to-coronary artery bypasses and their anti-ischemic effect has - for the first time - been recently demonstrated by our research group. The acute functional changes observed in response to temporary distal IMA balloon occlusion are expected to result in larger chronic structural adaptations of the IMA-to-coronary-artery connections when the distal IMA is permanently occluded. In contrast to the previously employed arteriogenic approaches in humans, the attractiveness of such an intervention lies in the potential durability of the effect.

In a first step, catheter-based IMA occlusion ought to be conceptually investigated in the setting of the less frequently grafted right IMA among patients with ischemia in the right coronary artery territory.

DETAILED DESCRIPTION:
Coronary artery disease and the benefit of bypasses:

Despite considerable advances in medicine, cardiovascular diseases remain the number one cause of death globally, primarily consequence of myocardial infarction (MI). Although widely used in stable CAD, percutaneous coronary intervention (PCI) has not been shown to reduce the incidence of myocardial infarction or death. In contrast, coronary artery bypass grafting (CABG) significantly reduced rates of death and myocardial infarction compared to PCI. Similarly, coronary collaterals exert a protective effect by providing an alternative source of blood flow to a myocardial territory potentially affected by an acute coronary occlusion. Coronary collaterals represent pre-existing inter-arterial anastomoses and as such are the natural counter-part of surgically created bypasses. Sufficient coronary collaterals have been shown to confer a significant benefit in terms of overall mortality and cardiovascular events. In this regard, the concept of augmenting coronary collateral function as an alternative treatment strategy to alter the course of CAD, as well as to control symptoms, is attractive.

Durable promotion of coronary collateral circulation:

While a multitude of interventions has been shown to be effective in collateral growth promotion, so far, the effect of current interventions is only temporary and therefore recurrent application is necessary to sustain the level of collaterals. However, before the advent of coronary artery bypass grafting, permanent augmentation of coronary collateral supply by a single structural modification has already been attempted. Bilateral ligation of the internal mammary arteries (IMA) was performed in CAD patients to alleviate angina pectoris and electrocardiographic (ECG) signs of ischemia. The prevalent in vivo function of natural IMA-to-coronary artery bypasses and their anti-ischemic effect has - for the first time - been recently demonstrated by our research group. Levels of collateral function and myocardial ischemia were determined during two coronary balloon occlusions, the first with, the second without distal IMA balloon occlusion. Coronary collateral function, was consistently increased in the presence vs the absence of distal ipsilateral IMA balloon occlusion. These findings were corroborated by the observed reduction in ischemia. Conversely, with distal contralateral IMA occlusion, collateral function and ECG signs of ischemia remained unchanged. The acute functional changes observed in response to temporary distal IMA balloon occlusion are expected to result in larger chronic structural adaptations of the IMA-to-coronary-artery connections when the distal IMA is permanently occluded. In contrast to the previously employed arteriogenic approaches in humans, the attractiveness of such an intervention lies in the potential durability of the effect.

In a first step, catheter-based IMA occlusion ought to be conceptually investigated in the setting of the less frequently grafted right IMA among patients with ischemia in the right coronary artery territory.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Referred for elective coronary angiography
* Written informed consent to participate in the study
* Significant stenosis of right coronary artery (FFR ≤0.80)

Exclusion Criteria:

* Acute coronary syndrome; unstable cardiopulmonary conditions, unstable angina pectoris
* Collateral flow index of right IMA <0.25
* Severe cardiac valve disease
* Congestive heart failure NYHA III-IV
* Prior coronary artery bypass surgery / prior cardiac surgery
* Coronary artery disease best treated by coronary artery bypass grafting
* Coronary artery disease unsuitable for intracoronary pressure measurements
* Prior Q-wave myocardial infarction in the vascular territory undergoing collateral function determination
* Severe renal or hepatic failure
* Women of childbearing age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in right coronary Collateral Flow Index (CFI) | Follow-up (week 6)
  Change from baseline in right coronary Collateral Flow Index (CFI) at follow-up (week 6) vs baseline

SECONDARY OUTCOMES:
Change from baseline in left coronary CFI | Follow-up (week 6)
  Change from baseline in left coronary CFI at follow-up (week 6) vs baseline
Change from baseline in intracoronary and surface ECG ST-segment shift during temporary right and left coronary balloon occlusion | Follow-up (week 6)
  Change from baseline in intracoronary and surface ECG ST-segment shift during temporary right and left coronary balloon occlusion at follow-up (week 6) vs baseline
Number of patients with angiographic visibility of right IMA-to-coronary anastomoses | Follow-up (week 6)
  Angiographic visibility of right IMA-to-coronary anastomoses at follow-up
Number of patients with catheter-based permanent right IMA occlusion | Baseline, Follow-up (week 6)

CONTACTS AND LOCATIONS:
Overall Officials: Seiler Christian, MD, Prof, Principal Investigator — Bern University Hospital
Locations (1):
- Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Stoller M, de Marchi SF, Seiler C. Function of natural internal mammary-to-coronary artery bypasses and its effect on myocardial ischemia. Circulation. 2014 Jun 24;129(25):2645-52. doi: 10.1161/CIRCULATIONAHA.114.008898. Epub 2014 Apr 17. PMID 24744276
- [Background] Moberg A. Anastomoses between extracardiac vessels and coronary arteries. II. Via internal mammary arteries. Post-mortem angiographic study. Acta Radiol Diagn (Stockh). 1967 May;6(3):263-72. doi: 10.1177/028418516700600306. No abstract available. PMID 6025072
- [Background] BLAIR CR, ROTH RF, ZINTEL HA. Measurement of coronary artery blood-flow following experimental ligation of the internal mammary artery. Ann Surg. 1960 Aug;152(2):325-9. doi: 10.1097/00000658-196008000-00018. No abstract available. PMID 13801236
- [Derived] Stoller M, Seiler C. Effect of Permanent Right Internal Mammary Artery Closure on Coronary Collateral Function and Myocardial Ischemia. Circ Cardiovasc Interv. 2017 Jun;10(6):e004990. doi: 10.1161/CIRCINTERVENTIONS.116.004990. PMID 28566292